CLINICAL TRIAL: NCT06452095
Title: RECLAIM: Recovering From COVID-19 Lingering Symptoms Adaptive Integrative Medicine Trial - Effect of Hyperbaric Oxygen Therapy for the Treatment of Post COVID Condition (RECLAIM-HBOT)
Brief Title: Recovering From COVID-19 Lingering Symptoms Adaptive Integrative Medicine Trial - Effect of Hyperbaric Oxygen Therapy for the Treatment of Post COVID Condition
Acronym: RECLAIM-HBOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-6203-HBOT
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Long COVID; Post Acute Sequelae of COVID-19; Post-COVID-19 Condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: RECLAIM is a Canada-wide phase ll/lll, prospective, adaptive randomized controlled platform trial that is intended to study various interventions for patients with long COVID. Interventional arms may be discontinued based on interim analysis results and new interventions may be selected and included as part of the platform as the trial progresses. As such, the protocol and consent documents are a modular design.
  The HBOT arm includes:
  * Master Protocol and informed consent documents: Contain information applicable to the whole platform.
  * HBOT Sub-Protocol: Contain additional information, specific to the HBOT interventional arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded to intervention in so far as the HBOT experience will be similar between treatment and sham arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): HBOT GROUP will have HBOT with 100% oxygen for 90 min, once daily, five times a week for 8 consecutive weeks. This will be given at a slightly higher pressure than normal air pressure (2 times regular air pressure)
  Interventions: Device: Hyperbaric Oxygen therapy
- Hyperbaric oxygen sham (Sham Comparator): CONTROL GROUP will have sham treatment, which will look and feel like HBOT, but will not have high enough oxygen concentration for any therapeutic or health benefit. Sham treatment with 21% oxygen (the amount of oxygen normally present in the air) for 90 min, once daily, five times a week for 8 consecutive weeks. This will be given at standard atmospheric pressure (1.03 ATA). The air pressure will vary slightly to mimic the feeling of HBOT.
  Interventions: Device: Hyperbaric Oxygen therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen therapy — The SECHRIST INDUSTRIES mono-place Hyperbaric Chambers OR Sigma Series mono-place Hyperbaric Chambers

SUMMARY:
The RECLAIM study platform will be used to explore whether the use of Hyperbaric Oxygen therapy (HBOT) improves the symptoms of post covid cognitive dysfunction.

Hyperbaric oxygen therapy is a well-established medical treatment. HBOT promotes healing by delivering a high concentration of oxygen into the body. This high level of oxygen has a number of known benefits, such as growth of new blood vessels, as well as regulating immune and inflammation responses. It helps protect the brain and other nervous tissue from inflammation. HBOT may also have antiviral effects.

Collectively, it has the potential to target the underlying mechanisms believed to play a critical role in the development of Long COVID.

Many individuals with Long COVID complain of fatigue, brain fog, muscle aches and other symptoms. There is evidence to suggest that these symptoms may be a problem with the blood vessels, resulting in abnormal delivery of oxygen to tissues. Thus, our group is investigating whether HBOT improves post-COVID cognitive dysfunction.

DETAILED DESCRIPTION:
This is a Sub-Protocol to the Core Clinical Study Protocol titled: REcovering from COVID19 Lingering symptoms Adaptive Integrative Medicine (RECLAIM),

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Positive COVID-19 test by nasopharyngeal swab RT-PCR (reverse transcription polymerase chain reaction) test, antibody or antigen tests at least 3 months prior to randomization; OR Presumed COVID-19 assessed by the site investigator (no positive COVID-19 test) with acute illness after October 15, 2019.
3. Patients should be treated with standard of care therapies (as discussed in the study manual) for at least 4 weeks prior to entry into trial.
4. Lingering COVID-19 symptoms beyond 3 months from onset of acute COVID and symptoms have lasted at least 2 months. The onset of COVID is considered the earliest of two dates: the date of positive test or the date of first symptoms;
5. Lingering symptoms from COVID-19 present at the time of randomization. "Lingering symptoms of Long COVID" must include self-reported cognitive dysfunction symptoms.
6. Female patients of childbearing potential (as assessed by the overseeing Investigator) who are sexually active must agree to practice true abstinence or use effective methods of contraception while on study treatment. Effective methods of contraception must be discussed and approved by the overseeing Investigator.
7. Must be able to provide informed consent and both willing and able to comply with study requirements.
8. A confirmed ability to travel to one of the three sites where HBOT or sham can be administered.

Exclusion Criteria:

1. Patients who had mechanical ventilation or extracorporeal membrane oxygen (ECMO) for COVID-19;
2. Current end-organ failure, organ transplantation, or current hospitalization in acute care hospital;
3. Contraindications to all of the study interventions;
4. Co-enrolment in another interventional trial (co-enrolment in an observational study is permitted);
5. Currently pregnant or breastfeeding.
6. Pneumothorax
7. Poorly controlled seizure disorder
8. Chronic sinusitis
9. Chronic or acute otitis media
10. Major ear drum trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Simple reaction time [SRT] task from the TestMyBrain (TMB) Digital Neuropsychology Toolkit | Baseline/Start of intervention to two months
  On-line survey tool
Verbal paired associates [VPA] task from the TestMyBrain (TMB) Digital Neuropsychology Toolkit | Baseline/Start of intervention to two months
  On-line survey tool

SECONDARY OUTCOMES:
Symptoms scale | Baseline/start of intervention weekly to 2 months, then once monthly to 6 months.
  Three point Likert scale assessing how bothersome symptoms are on a weekly basis for two months then monthly until end of study, as reported by the participant: to provide a granular, detailed picture of the symptom trajectory.
Symptom Checklist | Baseline/start of intervention to 1, 2 months 3 and 6 months
  Symptom Checklist (adapted from the De Paul Symptom Questionnaire (DSQ2), the World Health Organization Global COVID-19 Clinical Platform's Post COVID-19 CRF and the Symptom Burden Questionnaire for Long COVID): to track symptom trajectory.
Six Minute Walking Test (6MWT) with oximetry | Baseline/start of intervention and 2 months.
  Subjects walk as far as they can in six minutes while receiving maximum encouragement. It is simple to execute, inexpensive, standardized and gives a tangible measure of functional exercise capacity. It has been validated in many different populations. The 6MWT will be conducted according to American Thoracic Society standards.
SF-36 | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The self-administered SF-36 evaluates eight health concepts: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning-emotional, and mental health. Previous studies have used this instrument in many different populations and it takes approximately 15 minutes to complete.
TestMyBrain cognitive testing | Baseline/start of intervention to 1, 2 months 3 and 6 months
  TestMyBrain was developed as a tool to collect large, population-based samples for understanding the relationship between cognition, emotion, social functioning, and health. This test battery includes:
  TMB Verbal Paired Associates (Concrete), TMB Digit Span - Backward, TMB Digit Span - Forward, TMB Choice Reaction Time, TMB Simple Reaction Time, TMB Gradual Onset Continuous Performance Task. The test battery will take about 20 minutes to complete and will assess: verbal, episodic and working memory, attention, processing speed, basic psychomotor response speed, and cognitive control.
Post COVID19 functional status scale | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The post-COVID-19 functional status (PCFS) scale focuses on relevant aspects of daily life during follow-up after the infection. The scale is intended to help users become aware of current functional limitations in COVID-19 patients, whether or not as a result of the specific infection, and to objectively determine this degree of disability. The scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death), and covers the entire range of functional outcomes by focusing on limitations in usual duties/activities either at home or at work/study, as well as changes in lifestyle. The PCFS demonstrates good construct validity.
Reintegration to Normal Living Index (RNLI) | Baseline/start of intervention to 1, 2 months 3 and 6 months
  This short self-administered assessment tool will determine the degree to which participants reintegrate into normal social activities such as recreation, mobility in the community and interaction in family and other relationships. This tool has been validated in community living adults with mobility limitations.
The Fatigue Scale | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The Fatigue Scale was adapted from the De Paul Symptom Questionnaire (DSQ2)'s 38 questions assessing medical history of Myalgic Encephalitis/Chronic Fatigue Syndrome (ME/CFS), comorbidities, medications, impact on quality of life and daily activities, etc.
Brief Fatigue inventory | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The self-administered Brief Fatigue Inventory is composed of 9 items evaluated on a 10-point scale, assessing severity of fatigue and impact of fatigue on daily life. It takes approximately 2-3 minutes to complete.
Post-Exertional Malaise | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The self-administered DPEMQ is comprised of three sections assessing post-exertional malaise (PEM): (i) onset and triggers of PEM (9 questions), (ii) consequences and symptoms (14 questions), (iii) duration, recovery and pacing (7 questions).
Mental Health - General Anxiety Assessment Form (GAD-7) | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The GAD-7 is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. It is an easy-to-use, self-administered patient questionnaire that can be completed in minutes.
Mental Health - Patient Health Questionnaire (PHQ-9) | Baseline/start of intervention to 1, 2 months 3 and 6 months
  The PHQ-9 is a validated, multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It incorporates Diagnostic and Statistical Manual 1V (DSM-IV) depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The PHQ-9 is brief and useful in clinical practice.
Dyspnea | Baseline/start of intervention to 1, 2 months 3 and 6 months
  Assessed using the Borg Dyspnea scale. This short assessment tool assesses perceived shortness of breath on exertion using a 10 point scale as assessed by the patient.
Blood samples | Baseline/start of intervention and 2 months
  Blood samples will be used in correlative studies using advanced multi-omic and machine learning techniques to better understand our results so as to identify phenotypes that will benefit from specific therapies

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD, PhD, Study Director — University Health Network, Toronto; Rita Katznelson, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: Undecided